CLINICAL TRIAL: NCT01867762
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled, Efficacy and Safety Study of Inhaled JNJ 49095397 (RV568) in Subjects With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: An Effectiveness and Safety Study of Inhaled JNJ 49095397 (RV568) in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR101807; 49095397OPD2001 (Other: Janssen Research & Development, LLC); 2012-005184-27 (EudraCT Number)
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease; JNJ 49095397; RV568; Forced expiratory volume in one second; FEV1
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- JNJ 49095397 (Experimental)
  Interventions: Drug: JNJ 49095397
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ 49095397 — JNJ 49095397 400 microgram will be inhaled by participants once daily by using a dry powder inhaler for 12 weeks.
  Arms: JNJ 49095397
Drug: Placebo — Placebo will be inhaled by participants once daily by using a dry powder inhaler for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of JNJ 49095397 in participants with symptomatic moderate to severe chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This is a randomized (the study medication is assigned by chance), double-blind (neither physician nor participant knows the treatment that the participant receives), placebo-controlled (an inactive substance that is compared with a medication to test whether the medication has a real effect in a clinical study), multicenter, parallel-group (each group of participants will be treated at the same time) study. Approximately 200 participants will be randomly assigned to JNJ 49095397 or placebo in the ratio 1:1. The study consists of 3 phases: screening (3 weeks), double-blind treatment (12 weeks), and follow up (4 weeks). Safety evaluations will include assessment of adverse events, vital signs, physical examination, electrocardiograms, and clinical laboratory tests which will be monitored throughout the study. The total duration of the study for each participant will be approximately 19 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of non-child-bearing potential, Global Initiative for Chronic Obstructive Lung Disease (GOLD 2 or 3), forced expiratory volume in one second (FEV1) greater than or equal to 40 less than 80 percent predicted, FEV1/ forced vital capacity (FVC) ratio less than 0.7
* Clinical history of chronic bronchitis. Either two chronic obstructive pulmonary disease (COPD) exacerbations in past two years or ability to produce a spontaneous sputum sample, treated with long-acting beta-2 agonist (LABA)/ long-acting muscarinic antagonists (LAMA), with or without inhaled corticosteroids for at least 12 weeks prior to study entry
* Smoker or ex-smoker with at least a 10 pack-year history
* No COPD exacerbation that requires change in COPD maintenance medications during the screening period
* Not experienced a significant worsening of COPD based on clinical symptoms and by investigations during screening period

Exclusion Criteria:

* Has another pulmonary disease (eg, asthma) or an active infection (eg, tuberculosis)
* Has experienced life-threatening COPD (eg, requiring intensive care unit [ICU] admission, intubation, or long-term non-invasive ventilation). Short-term (less than five days), non-invasive ventilation during a hospitalization for an acute exacerbation of COPD is permitted, provided that non-invasive ventilation was not continued at home
* Has right heart failure or oxygen saturation less than 90 percent at rest on room air at screening or requires oxygen therapy on a daily basis for chronic hypoxemia (deficiency of oxygen in blood)
* History of significant disease or medical illness within 12 months prior to screening - Positive serology to human immunodeficiency virus (HIV)-1 or HIV-2, hepatitis B virus, or hepatitis C virus at screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2013-09-09 (Actual); Primary Completion 2014-08-06 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Prebronchodilator (preBD, before taking an inhaled bronchodilator) Percent-predicted Forced Expiratory Volume in one Second (FEV1) at Week 12 | Baseline (Week 0) to Week 12
  FEV1 is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.

SECONDARY OUTCOMES:
Change From Baseline in Postbronchodilator (postBD, after taking an inhaled bronchodilator) FEV1 at Week 12 | Baseline (Week 0) to Week 12
  FEV1 is the amount of air that can be exhaled in one second. FEV1 will be measured by spirometry. A positive change from baseline in FEV1 indicates improvement in lung function.
Change From Baseline in Weekly Average Number of Occasions in a day that Rescue Medication is Used at Week 12 | Baseline (Week 0) to Week 12
  Use of inhaled rescue medication (expressed as the number of occasions) taken on a schedule and/or for control of symptoms will be recorded twice daily.
Change From Baseline in EXAcerbations of Chronic Pulmonary Disease Tool-Respiratory Symptoms (E-RS) at Week 12 | Baseline (Week 0) to Week 12
  E-RS is an 11-items respiratory system scoring algorithm to assess the severity of respiratory symptoms in participants with chronic obstructive pulmonary disease (COPD). Each item has either 5 or 6 response options. Higher score indicates more severe COPD.
Change From Baseline in the Total Score of the St. George's Respiratory Questionnaire for COPD Patients (SGRQ-C) at Week 12 | Baseline (Week 0) to Week 12
  SGRQ-C is a 40-item questionnaire designed to measure health impairment in participants with COPD. SGRQ-C is divided into two components: 1) symptoms, 2) activity& impacts. Total SGRQ-C score ranges from 0 (best) and 100 (worst). Higher scores indicate greater health impairment.
Number of participants with adverse events | Up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (47):
- United States (6):
  - Phoenix, Arizona
  - St Louis, Missouri
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Spartanburg, South Carolina
- Belgium (5):
  - Antwerp
  - Brussels
  - Genk
  - Kortrijk
  - Leuven
- Canada (8):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Hamilton, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sainte-Foy, Quebec
  - Sherbrooke, Quebec
- Prague, Czechia
- Germany (6):
  - Berlin
  - Frankfurt
  - Großhansdorf
  - Hamburg
  - Lübeck
  - Mainz
- Hungary (4):
  - Budapest
  - Farkasgyepü
  - Mosonmagyaróvár
  - Szikszó
- Netherlands (5):
  - Eindhoven
  - Groningen
  - Rotterdam
  - Sittard / Geleen
  - Zwolle
- Poland (3):
  - Bialystok
  - Lodz
  - Wroclaw
- Bucharest, Romania
- Russia (3):
  - Barnaul
  - Moscow
  - Saint Petersburg
- United Kingdom (5):
  - Bristol
  - Dundee
  - Edinburgh
  - Glasgow
  - London